CLINICAL TRIAL: NCT02564575
Title: Phase 1 Evaluation of a Live Attenuated Human Parainfluenza Virus Type 3 Vectored Vaccine Candidate Expressing Ebolavirus Zaire Glycoprotein
Brief Title: Evaluating the Safety of and Immune Response to a Human Parainfluenza Virus Type 3 Ebola Virus Vaccine (HPIV3-EbovZ GP) in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CIR 305
Record Dates: First submitted 2015-09-29; First posted 2015-09-30 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2017-01

CONDITIONS: Hemorrhagic Fever, Ebola
Keywords: Ebolavirus
MeSH Terms: conditions — Hemorrhagic Fever, Ebola

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cohort 1 (Experimental): Participants will receive two doses, separated by 4-8 weeks, of approximately 10^6 PFU/mL of the HPIV3-EbovZ GP vaccine.
  Interventions: Biological: HPIV3-EbovZ GP Vaccine
- Cohort 2 (Experimental): Participants will receive two doses, separated by 4-8 weeks, of approximately 10^7 PFU/mL of the HPIV3-EbovZ GP vaccine.
  Interventions: Biological: HPIV3-EbovZ GP Vaccine

INTERVENTIONS:
Biological: HPIV3-EbovZ GP Vaccine — Administered intranasally by a VaxINator device

SUMMARY:
The purpose of this study is to evaluate the safety, infectivity, and immunogenicity of the HPIV3-EbovZ GP Ebola vaccine candidate in healthy adults.

DETAILED DESCRIPTION:
The ongoing Ebola virus outbreak in West Africa highlights the need for prevention and treatment strategies, as supportive therapy is currently the only treatment for Ebola virus disease. The purpose of this study is to evaluate the safety, infectivity, and immunogenicity of two doses of the HPIV3-EbovZ GP vaccine candidate administered intranasally in healthy adults.

This study will enroll healthy adults who have low pre-existing serum antibody titers to human parainfluenza virus type 3 (HPIV3). Participants will be enrolled sequentially in two cohorts. Cohort 1 will receive two doses of 10^6.0 PFU/mL of HPIV3-EbovZ GP, approximately 4-8 weeks apart. Cohort 2 will receive two doses of 10^7.0 PFU/mL of HPIV3-EbovZ GP, approximately 4-8 weeks apart.

Participants will be admitted to the inpatient unit 1 or 2 days before receiving their first dose of the vaccine. While in the inpatient unit, all participants will undergo a medical history review, physical examination, nasal wash, blood collection, pregnancy testing (for female participants), and pregnancy prevention counseling. Participants will be discharged from the inpatient unit on Day 7 or possibly later, depending on the results of participant's lab tests. An additional study visit will occur at Day 14.

On Day 26, participants will be readmitted to the inpatient unit, and they will receive their second dose of the vaccine on Day 28. Participants will undergo the same study procedures that occurred during the first inpatient stay, and they will be discharged on Day 35. Additional study visits will occur on Days 42, 56, 84, 112, 180, 270, and 360.

ELIGIBILITY:
Inclusion Criteria:

* Adult males and non-pregnant females between 18 years and 50 years of age inclusive. Children will not be recruited or enrolled in this study for safety considerations and because of the need for isolation.
* General good health, without significant medical illness, physical examination findings, or significant laboratory abnormalities as determined by the investigator.
* Low pre-existing serum antibody titers to HPIV3 (HAI titer less than or equal to 1:128).
* Agree to storage of blood specimens for future research.
* Available for the duration of the trial.
* Willingness to participate in the study as evidenced by signing the informed consent document.
* Female subjects of childbearing potential must agree to use effective birth control methods for the duration of the study (for example, pharmacologic contraceptives including oral, parenteral, subcutaneous and transcutaneous delivery; condoms with spermicide; diaphragm with spermicide; intrauterine device; abstinence from heterosexual intercourse; surgical sterilization). All female subjects will be considered being of childbearing potential except those who have undergone documented hysterectomy or bilateral oophorectomy, and those in whom menopause occurred at least 1 year prior to the study, confirmed by testing.
* Willingness to refrain from blood donation during the course of the study.
* Willingness to refrain from receiving other vaccines or investigational products during the first 4 months of the study after enrollment.

Exclusion Criteria:

* Pregnancy as determined by a positive human choriogonadotropin (beta-HCG) test.
* Currently breastfeeding.
* Evidence of clinically significant neurologic, cardiac, pulmonary, hepatic, rheumatologic, autoimmune, or renal disease by history, physical examination, and/or laboratory studies.
* History of intranasal pathology or evidence of structural abnormalities of the sinuses or nasal cavity upon examination.
* Behavioral or cognitive impairment or psychiatric disease that in the opinion of the investigator affects the ability of the subject to understand and cooperate with the study protocol.
* Positive urine drug toxicology test indicating narcotic use or history of dependency.
* Have medical, occupational, or family problems as a result of alcohol or illicit drug use during the past 12 months.
* Other condition that in the opinion of the investigator would jeopardize the safety or rights of a subject participating in the trial or would render the subject unable to comply with the protocol.
* History of anaphylaxis.
* Current diagnosis of asthma or reactive airway disease (within the past 2 years).
* Current history of allergic rhinitis requiring the use of medication.
* History of Bell's palsy.
* Positive ELISA and confirmatory test (e.g., Western blot or HIV-1/HIV-2 differentiation assay) for human immunodeficiency virus-1 (HIV-1).
* Positive ELISA and confirmatory test (e.g., PCR for virus) for hepatitis C virus (HCV).
* Positive hepatitis B virus surface antigen (HBsAg) by ELISA.
* Known immunodeficiency syndrome or history suggestive of impaired immune function.
* Use of corticosteroids (excluding topical preparations) or immunosuppressive drugs within 30 days prior to vaccination.
* Receipt of a live vaccine within 4 weeks or a killed vaccine within 2 weeks prior to study vaccination.
* History of asplenia.
* Body mass index (BMI) less than 18.5 or greater than 40.
* Receipt of blood or blood-derived products (including immunoglobulin) within 6 months prior to study vaccination.
* Current smoker unwilling to stop smoking for the duration of the inpatient study.

  * A current smoker includes anyone stating they currently smoke any amount of a tobacco product.
  * The decision to exclude a potential subject is determined by medical history and a clinician's clinical judgment based on the physical examination.
  * After admission to the unit, nicotine patches will be provided to current smokers who request them for the inpatient portion of the study.
* Travel to Liberia, Sierra Leone or Guinea in the last 12 months or are intending to travel to an Ebola endemic region during the study period.
* Receipt of another investigational vaccine or drug within 30 days prior to study vaccination.
* Previous receipt of an investigational Ebola or Marburg virus vaccine, a chimpanzee adenovirus, or HPIV vectored vaccine or any other investigational vaccine likely to impact on interpretation of the trial data.
* Individuals with current or past (in the last 4 weeks) use of intranasal medications (including steroids, decongestants, or hormonal medications) or who have plans to use them within 28 days of study vaccination.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-08; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Frequency of vaccine-related reactogenicity events | Measured through Day 56
Number of vaccinees infected with HPIV3-EbovZ GP vaccine virus when given at 10^6.0 or 10^7.0 PFU | Measured through Day 360
  Infection is defined as the recovery of vaccine virus from nasal wash, and/or the detection of virus in nasal wash by rRT-PCR, and/or a ≥4-fold rise in serum antibody titer to ebolavirus GP or HPIV3.
The titer of vaccine virus recovered from nasal wash specimens obtained from each recipient | Measured through Day 360
Number of days vaccine virus was shed, measured by plaque titration and rRT-PCR | Measured through Day 360

SECONDARY OUTCOMES:
Development of serum antibody to the EbovZ-GP | Measured through Day 360

CONTACTS AND LOCATIONS:
Overall Officials: Kawsar Talaat, MD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Center for Immunization Research (CIR), Johns Hopkins Bloomberg School of Public Health (JHBSPH), Baltimore, Maryland, United States